CLINICAL TRIAL: NCT04967235
Title: Dance Therapy as an Alternative for Cardiac Rehabilitation in Women Population: Autonomic and Hemodynamic Acute Responses - A Crossover Clinical Trial
Brief Title: Dance Therapy as an Alternative for Cardiac Rehabilitation in Women Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Responsible Party: Principal Investigator, Luiz Carlos Marques Vanderlei, PhD, Universidade Estadual Paulista Júlio de Mesquita Filho
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 79786017.5.0000.5402
Record Dates: First submitted 2021-07-13; First posted 2021-07-19 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Cardiac Risk Factors; Cardiovascular Diseases
Keywords: Cardiac Rehabilitation; Dance Therapy; Cardiac Risk Factors; Autonomic Nervous System; Heart Rate
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: The study consists of one group of women who will be submitted to one dance-based cardiac rehabilitation session and after that will be submitted to one conventional exercise-based cardiac rehabilitation session
Who Masked: Investigator, Outcomes Assessor
Masking Description: The researcher performing the heart rate variability and heart rate recovery data filtering will be blinded, and the researcher performing the data analysis will also be blinded. All data will be handled in a coded datasheet and all volunteer's names will be replaced by a confidential ID.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Exercise-based Cardiac Rehabilitation (Active Comparator): This interventional arm consists of a conventional exercise-based cardiac rehabilitation, composed of initial rest, warm-up, treadmill aerobic exercise, orthostatic passive recovery, and supine passive recovery.
  Interventions: Other: Conventional Exercise-based Cardiac Rehabilitation Session
- Dance-Based Cardiac Rehabilitation (Experimental): This interventional arm consists of a new dance-based cardiac rehabilitation, composed of initial rest, warm-up, dance therapy, orthostatic passive recovery and supine passive recovery.
  Interventions: Other: Dance-based Cardiac Rehabilitation Session

INTERVENTIONS:
Other: Conventional Exercise-based Cardiac Rehabilitation Session — This session will be composed of:
  I.10 minutes of initial rest in the supine position; II. 15 minutes of warm-up through stretching and global exercises; III. 30 minutes of treadmill aerobic exercise at an intensity of 60-80% of the heart rate reserve for those without diabetes Mellitus and 40-70% of the heart rate reserve for those diagnosed with diabetes mellitus; IV. 1 minute passive recovery in orthostatic position; V. 30 minutes of passive recovery in the supine position.
  Arms: Conventional Exercise-based Cardiac Rehabilitation
Other: Dance-based Cardiac Rehabilitation Session — I.10 minutes of initial rest in the supine position; II. 15 minutes of warm-up through stretching and global exercises; III. 30 minutes of dance therapy. The intensity of the choreography will be set at the same range as the conventional exercise-based session. (60-80% of the heart rate reserve for those without diabetes Mellitus and 40-70% of the heart rate reserve for those diagnosed with diabetes mellitus); IV. 1 minute passive recovery in orthostatic position; V. 30 minutes of passive recovery in the supine position.
  Arms: Dance-Based Cardiac Rehabilitation

SUMMARY:
This research project aims to investigate the acute effects of a dance-based cardiac rehabilitation session in the cardiovascular system and autonomic modulation of women with cardiac risk factors. Also, as a secondary outcome, to compare the cardiovascular and autonomic responses of the dance-based session to a conventional exercise-based session.

ELIGIBILITY:
Inclusion Criteria:

* Hemodynamically stable
* Previously attending exercise-based cardiac rehabilitation and dance classes for at least 3 months
* Do not present orthopedics or neurologic impairments that could preclude the execution of dance movements
* To be previously diagnosed with at least one of the following cardiac risk factors:

  1. Age ≥ 55 years
  2. Family history: Known myocardial infarction, coronary revascularization, or sudden death in the first-degree relatives before 55 years in male or 65 years in female relatives
  3. Hypertension: values of systolic blood pressure (SBP) equal to or higher than 140 mmHg and/or values of diastolic blood pressure (DBP) equal to or higher than 90 mmHg, or daily use of antihypertensive drugs
  4. Dyslipidemia: values of low-density lipoprotein (LDL) ≥ 130 mg.dL-1, or values of high-density lipoprotein (HDL) < 40 mg.dL-1, or daily use of lipid-lowering drugs
  5. Obesity: body mass index ≥ 30 Kg.m-2
  6. Cigarette smoking: former smokers for more than six months
  7. Diabetes Mellitus: fasting blood glucose level ≥ 100 mg.dL-1
  8. Physically inactivity: the volunteer will be considered physically inactivity when classified as "sedentary" or "irregularly active A or B" by the International Physical Activity Questionnaire (IPAQ)
  9. Stress: the presence of stress will be evaluated by the Lipp's Stress Symptoms Inventory (LSSI), and the classifications "alert", "resistance", and "exhaustion" will be considered

Exclusion Criteria:

* Volunteers who present errors superior to 5% in the RR intervals time series
* Volunteers who do not attend all study phases

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Heart Rate | Acute evaluation during interventions
  The heart rate will be collected using a heart rate monitor (Polar RS800CX - Polar Electro, Kempele, Finland). The data will be assessed at the 5th minute of initial rest, and at the 1st, 2nd, 3rd, 5th, 10th, 20th, and 30th minutes of passive recovery in supine position.
Blood Pressure | Acute evaluation during interventions
  Evaluated indirectly by an experienced physiotherapist using a stethoscope and a sphygmomanometer. This data will be assessed at he 5th minute of initial rest, and at the 1st, 2nd, 3rd, 5th, 10th, 20th, and 30th minutes of passive recovery in supine position.
Peripheral oxygen saturation | Acute evaluation during interventions
  Evaluated through a pulse oximeter (Mindray PM-50 Pulse Oximeter, China). This data will be assessed at he 5th minute of initial rest, and at the 1st, 2nd, 3rd, 5th, 10th, 20th, and 30th minutes of passive recovery in supine position.
Respiratory Rate | Acute evaluation during interventions
  Evaluated by an experienced and independent researcher that will count the number of respiratory incursions within one minute, without the volunteer noticing this procedure. This data will be assessed at he 5th minute of initial rest, and at the 1st, 2nd, 3rd, 5th, 10th, 20th, and 30th minutes of passive recovery in supine position.
Autonomic Modulation - rMSSD index | Acute evaluation during interventions
  The data for this evaluation will be collected using a heart rate monitor that registers the heart rate beat by beat and provides information regarding the RR intervals. This data will be analyzed in the following time sections: 5th to 10th min of initial rest, from the 5th to the 25th minute of resistance phase (treadmill exercise and dance therapy), and from the beginning to the end of the supine recovery phase. The rMSSD index corresponds to the root-mean square of differences between adjacent normal RR intervals in a time interval, expressed in milliseconds.
Autonomic Modulation - SDNN index | Acute evaluation during interventions
  The data for this evaluation will be collected using a heart rate monitor that registers the heart rate beat by beat and provides information regarding the RR intervals. This data will be analyzed in the following time sections: 5th to 10th min of initial rest, from the 5th to the 25th minute of resistance phase (treadmill exercise and dance therapy), and from the beginning to the end of the supine recovery phase. The SDNN index corresponds to the standard deviation of all normal RR intervals recorded in a time interval, expressed in milliseconds
Autonomic Modulation - LF index | Acute evaluation during interventions
  The data for this evaluation will be collected using a heart rate monitor that registers the heart rate beat by beat and provides information regarding the RR intervals. This data will be analyzed in the following time sections: 5th to 10th min of initial rest, from the 5th to the 25th minute of resistance phase (treadmill exercise and dance therapy), and from the beginning to the end of the supine recovery phase.The LF index is the low-frequency component of the oscillatory components of heart rate variability, and ranges from 0.04 to 0.15 Hz.
Autonomic Modulation - HF index | Acute evaluation during interventions
  The data for this evaluation will be collected using a heart rate monitor that registers the heart rate beat by beat and provides information regarding the RR intervals. This data will be analyzed in the following time sections: 5th to 10th min of initial rest, from the 5th to the 25th minute of resistance phase (treadmill exercise and dance therapy), and from the beginning to the end of the supine recovery phase. The HF index is the high-frequency component of the oscillatory components of heart rate variability, and ranges from 0.15 to 0.4 Hz.
Autonomic Modulation - TINN index | Acute evaluation during interventions
  The data for this evaluation will be collected using a heart rate monitor that registers the heart rate beat by beat and provides information regarding the RR intervals. This data will be analyzed in the following time sections: 5th to 10th min of initial rest, from the 5th to the 25th minute of resistance phase (treadmill exercise and dance therapy), and from the beginning to the end of the supine recovery phase. extracted from the density histogram constructed with all normal RR intervals, where the x-axis contains the RR intervals length, and the y-axis contains the frequency of occurrence of the RR intervals. The measure of the histogram base corresponds to the TINN index.
Autonomic Modulation - RRtri index | Acute evaluation during interventions
  The data for this evaluation will be collected using a heart rate monitor that registers the heart rate beat by beat and provides information regarding the RR intervals. This data will be analyzed in the following time sections: 5th to 10th min of initial rest, from the 5th to the 25th minute of resistance phase (treadmill exercise and dance therapy), and from the beginning to the end of the supine recovery phase. Extracted from the density histogram constructed with all normal RR intervals, where the x-axis contains the RR intervals length, and the y-axis contains the frequency of occurrence of the RR intervals. The ratio between the histogram area and the modal frequency corresponds to the RRtri index
Autonomic Modulation - SD1 index | Acute evaluation during interventions
  The data for this evaluation will be collected using a heart rate monitor that registers the heart rate beat by beat and provides information regarding the RR intervals. This data will be analyzed in the following time sections: 5th to 10th min of initial rest, from the 5th to the 25th minute of resistance phase (treadmill exercise and dance therapy), and from the beginning to the end of the supine recovery phase. The SD1 index corresponds to the dispersion of points perpendicular to the line of identity of the ellipse obtained from the Poincaré plot. Expressed in milliseconds.
Autonomic Modulation - SD2 index | Acute evaluation during interventions
  The data for this evaluation will be collected using a heart rate monitor that registers the heart rate beat by beat and provides information regarding the RR intervals. This data will be analyzed in the following time sections: 5th to 10th min of initial rest, from the 5th to the 25th minute of resistance phase (treadmill exercise and dance therapy), and from the beginning to the end of the supine recovery phase. The SD2 index corresponds to the dispersion of points along the line of identity of the ellipse obtained from the Poincaré plot. Expressed in milliseconds.
Autonomic Modulation - Recurrence rate | Acute evaluation during interventions
  The data for this evaluation will be collected using a heart rate monitor that registers the heart rate beat by beat and provides information regarding the RR intervals. This data will be analyzed in the following time sections: 5th to 10th min of initial rest, from the 5th to the 25th minute of resistance phase (treadmill exercise and dance therapy), and from the beginning to the end of the supine recovery phase. Extracted from the graph reconstruction of the spatial trajectory of the RR interval time series, the recurrence rate corresponds to the ratio of all recurrence states to all possible states.
Autonomic Modulation - Determinism | Acute evaluation during interventions
  The data for this evaluation will be collected using a heart rate monitor that registers the heart rate beat by beat and provides information regarding the RR intervals. This data will be analyzed in the following time sections: 5th to 10th min of initial rest, from the 5th to the 25th minute of resistance phase (treadmill exercise and dance therapy), and from the beginning to the end of the supine recovery phase. Extracted from the graph reconstruction of the spatial trajectory of the RR interval time series, the determinism corresponds to the ratio of recurrence points forming diagonal to all recurrence points.
Autonomic Modulation - Sample Entropy | Acute evaluation during interventions
  The data for this evaluation will be collected using a heart rate monitor that registers the heart rate beat by beat and provides information regarding the RR intervals. This data will be analyzed in the following time sections: 5th to 10th min of initial rest, from the 5th to the 25th minute of resistance phase (treadmill exercise and dance therapy), and from the beginning to the end of the supine recovery phase. Defined as the conditional probability that two sequences similar for n points remain similar at the next point, which indicates the series complexity.
Autonomic Modulation - Approximate Entropy | Acute evaluation during interventions
  The data for this evaluation will be collected using a heart rate monitor that registers the heart rate beat by beat and provides information regarding the RR intervals. This data will be analyzed in the following time sections: 5th to 10th min of initial rest, from the 5th to the 25th minute of resistance phase (treadmill exercise and dance therapy), and from the beginning to the end of the supine recovery phase. Measure the complexity of the series by examining the frequency in which similar epochs occurs.
Autonomic Modulation - Detrended fluctuation analysis (DFA) | Acute evaluation during interventions
  The data for this evaluation will be collected using a heart rate monitor that registers the heart rate beat by beat and provides information regarding the RR intervals. This data will be analyzed in the following time sections: 5th to 10th min of initial rest, from the 5th to the 25th minute of resistance phase (treadmill exercise and dance therapy), and from the beginning to the end of the supine recovery phase. Will be considered the DFA-total, the short-term alpha correlations - considering correlations from 4 to 11 RR intervals, and the long-term alpha correlations - considering 11 to 64 RR intervals.
Autonomic Modulation - Symbolic Analysis | Acute evaluation during interventions
  The data for this evaluation will be collected using a heart rate monitor that registers the heart rate beat by beat and provides information regarding the RR intervals. This data will be analyzed in the following time sections: 5th to 10th min of initial rest, from the 5th to the 25th minute of resistance phase (treadmill exercise and dance therapy), and from the beginning to the end of the supine recovery phase. This analysis indicates the quantity and type of variation between 3 consecutive RR intervals, classifying them in the following families: 0V (no variation), 1V (one variation), 2LV (two equal variations), and 2LV (two different variations. Also, will be analyzed the Shannon Entropy that is calculated by quantifying the frequency in which each family appears and summing the relative frequencies weighted by the logarithm of the inverse of the relative frequencies.

SECONDARY OUTCOMES:
Heart rate recovery of 1 minute | Acute evaluation during interventions
  The heart rate will be collected using a heart rate monitor (Polar RS800CX - Polar Electro, Kempele, Finland). The heart rate recovery of 1 minute (HRR1) will be calculated considering the following formula: HRR1 = HRpeak - HR1, where HRpeak will be determined by the mean of the last five beats registered at the resistance phase, and HR1 will be determined by the mean of the four beats around the heart rate registered exactly after one minute of recovery, two beats before and two beats after this value. This data will be extracted from the 1 minute orthostatic recovery.
30-seconds rMSSD | Acute evaluation during interventions
  The data for this evaluation will be collected using a heart rate monitor that registers the heart rate beat by beat and provides information regarding the RR intervals. This index will be calculated in the last 30 seconds of the resistance phase (treadmill exercise and dance therapy), and during the one minute of orthostatic passive recovery after the resistance phase.

CONTACTS AND LOCATIONS:
Overall Officials: Luiz Carlos M Vanderlei, PhD, Principal Investigator — Universidade Estadual Paulista "Julho de Mesquita Filho" (UNESP)
Locations (1):
- Universidade Estadual Paulista Júlio de Mesquita Filho, Presidente Prudente, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lucas Neves Silva JP, de Avila Soares JC, Lopez Laurino MJ, Ribeiro F, de Lima Gervazoni N, Spinardi Alves BI, Carvalho Novaes Moreira E, Marques Vanderlei LC, Modolo Regueiro Lorenconi R. Comparison of Nonlinear Dynamics of Heart Rate Variability Between Conventional Cardiac Rehabilitation and Dance-Based Therapy: A Non-Randomized Crossover Clinical Trial. J Dance Med Sci. 2025 Feb 19:1089313X251316672. doi: 10.1177/1089313X251316672. Online ahead of print. PMID 39968942